CLINICAL TRIAL: NCT03762967
Title: Efficiency Evaluation of Adipose-Derived Adult Stromal Vascular Cells in Patients With Spermatogenesis Disorders.
Brief Title: Autologous Adipose-Derived Adult Stromal Vascular Cell Administration for Male Patients With Infertility
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: State-Financed Health Facility "Samara Regional Medical Center Dinasty" (Other)
Responsible Party: Principal Investigator, Volchkov Stanislav, Deputy director, Quality assurance director, State-Financed Health Facility "Samara Regional Medical Center Dinasty"
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 23032018
Record Dates: First submitted 2018-11-27; First posted 2018-12-04 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Azoospermia; Oligozoospermia
Keywords: Autologous Stem Cell; Male infertility; Adipose-Derived stem cell; Azoospermia; Oligospermia
MeSH Terms: conditions — Azoospermia; Oligospermia; Infertility, Male | interventions — Standard of Care; Diet, Healthy

STUDY DESIGN:
Intervention Model Description: The study consist 40 patients in 4 groups. Two working groups and two control groups. Each group consist 10 Males.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Lipoaspiration and SVF introduction I. (Experimental): Patients with azoospermia that introduce with standard treatment and Lipoaspiration and SVF introduction.
  Interventions: Biological: Lipoaspiration and SVF introduction.; Drug: Standard therapy.
- Standard therapy I. (Active Comparator): Patients with azoospermia that introduce with Standard therapy only.
  Interventions: Drug: Standard therapy.
- Lipoaspiration and SVF introduction II (Experimental): Patients with oligospermia that introduce with standard treatment and Lipoaspiration and SVF introduction.
  Interventions: Biological: Lipoaspiration and SVF introduction.; Drug: Standard therapy.
- Standard therapy II. (Active Comparator): Patients with oligospermia that introduce with Standard therapy only.
  Interventions: Drug: Standard therapy.

INTERVENTIONS:
Biological: Lipoaspiration and SVF introduction. — Lipoaspiration, isolation of SVF and introduction into testis Interstitium.
  Arms: Lipoaspiration and SVF introduction I.; Lipoaspiration and SVF introduction II
Drug: Standard therapy. — Standard therapy include to give up bad habits, to establish a healthy diet, to eliminate excessive physical exertion. eliminate. In the case of endocrine disorders, hormone therapy is prescribed.
  Other Names: healthy diet, physical exertion eliminate. hormone therapy.

SUMMARY:
Severe Oligospermia (oligozoospermia) refer to semen with a low concentration of sperm and is a common finding in male infertility. Often semen with a decreased sperm concentration may also show significant abnormalities in sperm morphology and motility that affect Male fertility. The purpose of this study is to assess the ability of Autologous Adipose-Derived Adult Stromal Vascular Fraction (SVF) cells to stimulate Sertoli and spermatogonia cells and affect male fertility.

DETAILED DESCRIPTION:
This is an open-label study to evaluate efficiency of administration of Autologous Adipose-Derived Adult Stromal Vascular Fraction (SVF) in the testis in patients with oligospermia and azoospermia.

Forty men with several form oligozoospermia and azoospermia will be recruited for the study. 20 patients with same diagnosis served as a control with standard medications.Other patients -10 with oligospermia and 10 with azoospermia will receive standard medication and SVF injections.

The diagnosis of Azoospermia (Oligospermia) will be established on the basis of two and more semen analysis evaluations done at separate occasions and detailed history taking, physical examination and investigations (blood tests include hormon levels as testosteron. follicle stimulating hormone (FSH), luteinizing hormone (LH). karyotyping and testosterone levels, and may include testicular biopsy or transrectal ultrasound if indicated.

This study affect only Pretesticular and Testicular forms, without chromosomal aberration. SVF can produce a lot of cytokines ( as EGF, FGF, NGF, PDGF, VEGF, IGF, GMCSF, GCSF, TGF, Erythropoetin, TPO, BMP, HGF, GDF, Neurotrophins, MSF, SGF, GDF and growth factors) moreover the microvesicles and exosomes released by this cells can prevent cells from apoptosis and stimulate regenerative process of surrounding tissues and cells.

SVF will be transplanted by an andrological surgeon through a standard surgical approach. Subjects will be monitored frequently for a total of one year after cell injection.

ELIGIBILITY:
Inclusion Criteria:

* idiopathic oligozoospermia (spermatozoid number <2x10^6/mL) - 10 patients
* cryptozoospermia/azoospermia - 10 patients

Exclusion Criteria:

* age before 18 or after 60 years old
* heart insufficiency. stroke (during 1 year)
* anemia
* blood disease
* pelvis bone trauma
* chronic diseases in decompensation stage
* skin diseases
* tuberculosis
* hyperprolactinaemia
* hyper or hypothyreosis
* obstructive zoospermia
* sperm stimulating hormone therapy
* Men with previous surgery in testis
* Men with infectious genital diseases and anatomical abnormalities of the genital tract
* Those with major medical problems such as malignancy, hepatitis B . C, etc. HIV
* Chromosomal aberration (e.g. Y microdeletion, trisomy….)

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-03-12 (Actual); Primary Completion 2020-12-30 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
sperm concentration in ejaculate | 1, 2, 3 month
  Sperm quantity and quality will be evaluated with automatic sperm cout analyzer a month, two and three after injection of SVF. Total measures - 3.
Spermatozoa in testicular biopsy | 3 month
  Testicular sperm aspiration (TESA) will be performed after 3 month after SVF injection.

SECONDARY OUTCOMES:
Testosterone | 3 month
  Testosterone will be measured a three month after injection of SVF.
Inhibin-B | 3 month
  Inhibin-B will be measured a three month after injection of SVF.
Follicle stimulating hormone (FSH) | 3 month
  Follicle stimulating hormone will be measured a three month after injection of SVF.

CONTACTS AND LOCATIONS:
Overall Officials: Olga Tyumina, M.D. P.h.D., Study Chair — Medical Centre Dinasty
Locations (1):
- Medical Centre Dinasty, Samara, Russia